CLINICAL TRIAL: NCT01737073
Title: Comprehensive Opioid Management in Patient Aligned Care Teams (COMPACT)
Brief Title: Comprehensive Opioid Management in Patient Aligned Care Teams
Acronym: COMPACT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was unable to overcome IT and contracting barriers which prevented the study's data collection system from being implemented.
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: CRE 12-006; NCT02508285 (obsolete NCT alias)
Record Dates: First submitted 2012-11-26; First posted 2012-11-29 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Chronic Pain
Keywords: chronic pain; opioid; cognitive behavior therapy
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- IVR self management (Experimental): cognitive behavioral based self management training for chronic pain delivered by interactive voice response (IVR)
  Interventions: Behavioral: IVR self-management
- Opioid monitoring (Experimental): monthly interactive voice response (IVR) monitoring of prescription opioid use with feedback to the prescribing physician
  Interventions: Behavioral: Opioid monitoring
- IVR self management plus opioid monitoring (Experimental): Cognitive behavioral based self management training for chronic pain delivered by IVR plus monthly IVR monitoring of prescription opioid use with feedback to the prescribing physician
  Interventions: Behavioral: IVR self-management; Behavioral: Opioid monitoring
- Enhanced usual care (Other): Weekly automated wellness tips via IVR
  Interventions: Other: Enhanced usual care

INTERVENTIONS:
Behavioral: IVR self-management — A course of self-management training that includes 12 education and self-management skill modules presented over 12 consecutive weeks. Participants will be asked to practice each skill daily and report via IVR on their completion of the daily skill practice. They will receive a 10 minute call each week from a nurse care manager to discuss their weekly progress.
  Arms: IVR self management; IVR self management plus opioid monitoring
Behavioral: Opioid monitoring — Monthly automated monitoring of prescription opioid use including pain relief, physical activity, pain-related interference, mood, adverse effects, adherence and satisfaction with treatment.
  Arms: IVR self management plus opioid monitoring; Opioid monitoring
Other: Enhanced usual care — Weekly automated wellness tip and usual clinical care
  Arms: Enhanced usual care

SUMMARY:
This study will enroll Veterans with chronic pain who have been receiving opioid medications (like methadone, percocet, oxycontin) on a regular basis for at least 3 months to treat their pain. The purpose of this study is to understand if two automated interventions that are delivered by phone can improve the safe and effective use of opioid medications and the physical functioning of Veterans with chronic pain who take opioid medications. One intervention, opioid monitoring, will include monthly automated calls to the enrolled Veteran to ask questions about their use of the opioid medications, pain relief, side effects, effect of pain on physical activity and mood and satisfaction with pain care. The other intervention, skills training, includes learning pain management skills using automated calls and a self-help book with weekly feedback calls from a nurse. Veterans who are enrolled in this study will be randomly assigned (by chance, like a flip of a coin) to receive either opioid monitoring only, self-management only, self-management plus opioid monitoring or a weekly automated phone call with wellness tips. Everyone enrolled in the study will complete questionnaires about their pain and other pain-related information at the beginning of the trial, after the interventions are completed 12 weeks later, and 3 and 6 months after treatment ends.

DETAILED DESCRIPTION:
The objectives of the study are to: 1) test the effectiveness of an automated intervention system called COMPACT for improving pain-relevant outcomes including physical functioning and pain intensity; 2) determine whether opioid monitoring promotes guideline concordant care; and 3) examine key components of the intervention process to inform future implementation.

This study is a randomized, controlled, multi-site, factorial design trial of a technology supported treatment program called COMPACT relative to enhanced usual care (EUC) in the PACT setting. Participants will include 380 Veterans receiving chronic opioid therapy (COT) and reporting chronic musculoskeletal pain of at least moderate severity. Outcomes of interest include pain-related physical functioning, pain intensity, presence of guideline concordant care practices, and provider satisfaction. Enrolled participants will be randomized to receive COMPACT treatment or EUC. At baseline, 12 weeks (post-treatment), 24 weeks (follow-up) and 36 weeks (follow-up) all participants will undergo an opioid risk evaluation and assessment of all outcome variables. Participants randomized to COMPACT treatment will received interactive voice response (IVR)-based pain self management training and monthly opioid risk monitoring. Throughout treatment COMPACT participants will undergo automated monthly opioid risk monitoring and collection of patient reported opioid use, pain intensity, physical functioning, emotional functioning and quality of life data. Monthly opioid risk monitoring information will be made available to PACT clinicians via automatic entry into CPRS prior to a scheduled opioid renewal appointment. Participants in the EUC condition will undergo assessment of outcome variables and opioid risk assessment at 12-, 24- and 36-weeks post baseline only; they will not receive treatment or opioid monitoring.

ELIGIBILITY:
Inclusion Criteria:

* presence of at least moderate musculoskeletal diagnosis pain (i.e., pain scores of 4 as measured by the Numeric Rating Scale) for a period of 3 months. Musculoskeletal diagnosis is a cluster of disorders including:

  * low back and spine conditions
  * osteoarthritis
  * nerve compression
  * other inflammatory and degenerative disorders
* receipt of chronic opioid therapy [90 continuous days out of any 104 day period in the prior 12 month]
* ability to participate safely in the walking portion of the intervention as evidenced by patient-reported ability to walk at one block
* availability of a land line or cellular telephone

Exclusion Criteria:

* active psychosis or suicidality that could impair participation, identified using validated measures in the baseline screener
* life threatening or acute medical condition that could impair participation
* dementia defined by a score of 20 or greater on the St. Louis University Mental Status in the baseline screener
* any sensory deficits that would impair participation (e.g., hearing loss to a degree that telephone usage is not possible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory | Post-treatment (12 weeks post baseline)

SECONDARY OUTCOMES:
Concordance with opioid treatment practice guidelines | Post-treatment
  Evaluation of the effect of the OM intervention on providers' concordance with VA/DoD chronic opioid treatment practice guidelines will be a quality score (scale 0 - 8) that represents the number of practices out of eight key practices to which providers adhered at the 12 weeks follow up. The eight key practices considered are: use of UDS, contra-indicated co-prescription, non-medication treatments, no psychiatric at risk/SUD, acetaminophen over-prescription, risky sedative co-prescription, bowel regimen and serious adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Alicia A. Heapy, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No